CLINICAL TRIAL: NCT05043012
Title: Diagnostic Performance Of Non-Endorectal Coil Multiparametric Magnetic Resonance Imaging Of Prostate With Flexible AIR Coil (DoNEMAC Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1044; NCI-2021-09414 (Registry Identifier: CTRP (Clinical Trial Reporting Program)
Record Dates: First submitted 2021-08-24; First posted 2021-09-13 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): will have an mpMRI scan with a flexible AIR coil.
  Interventions: Device: flexible AIR coil
- Group 2 (Experimental): will have an mpMRI scan with an endorectal coil
  Interventions: Device: endorectal coi

INTERVENTIONS:
Device: flexible AIR coil — mpMRI scan
  Arms: Group 1
Device: endorectal coi — mpMRI scan
  Arms: Group 2

SUMMARY:
Multiparametric MRI (mpMRI) of the prostate is an important tool for diagnosis of clinically significant prostate cancer (csPCa) in men with an elevated serum prostate specific antigen, which can decrease the rate of unnecessary biopsies and reduce the incidence of over-diagnosis of non-csPCa. Furthermore, there is evidence that MRI is more accurate in detecting high-grade (Gleason grade group ≥3) versus low grade cancers (Gleason grade group <2) and therefore may serve as a useful adjunct to prostate-specific antigen (PSA) testing, digital rectal examination, and prostatic biopsy to detect cancers that require definitive treatment as opposed to active surveillance. Many investigators, including our group, have shown the utility of preoperative mpMRI to assess the local extent of prostate cancer and for surgical planning.

DETAILED DESCRIPTION:
Primary Objective:

To compare the detection rate of Gleason Group grade ≥ 2 disease in patients with intermediate and high-risk prostate cancer who undergo ERC mpMRI (Group 1: Control) versus patients who undergo non-ERC mpMRI with flexible AIR coil technology (Group 2: Experimental).

Secondary Objective:

1. To compare the scanning time and room time in Group 1 versus Group 2.
2. To compare patient-reported outcome at the end of the MRI test in Group 1 versus Group 2 through testing morbidities index (TMI).
3. To determine the impact of mpMRI on treatment planning for men with intermediate and high-risk prostate cancer and compare management impact in Group 1 versus Group 2
4. To compare the detection rate of T3 disease on MRI (confirmed by histopathology) at prostatectomy between Group 1 versus Group 2.

ELIGIBILITY:
Inclusion Criteria:

* Male, Age ≥ 18
* Untreated, biopsy-proven with intermediate and high-risk (Gleason group grade >/=2) adenocarcinoma of the prostate
* Patient is being considered for curative-intent treatment with radical prostatectomy within 6 months following mpMRI
* Patient has provided written informed consent for participation in this trial
* Patient should be eligible for scanning at 3 T magnet

Exclusion Criteria:

* Low-risk adenocarcinoma of prostate
* Patient has had any prior therapy for prostate cancer
* A history of other active malignancy within the last 2 years
* Prostate cancer with significant sarcomatoid or spindle cell or neuroendocrine small cell components
* Cardiac pacemaker
* Orthopedic hardware in the pelvis and spine.
* Claustrophobia and/or receiving anesthesia
* Contraindication for endorectal coil such as rectal bleeding, severe anal fissures or hemorrhoids, anal/rectal surgery, and lack of rectum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
To correlate the detection rate of Gleason Group grade ≥ 2 disease in patients with intermediate and high-risk prostate cancer who undergo ERC mpMRI | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tharakeswara Bathala, MBBS,MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org